CLINICAL TRIAL: NCT03500887
Title: A Pilot Study to Investigate Whether Intragastric Pressure During Food Intake Can be Measured Using an Intragastric Bag in Healthy Volunteers
Brief Title: Monitoring Stomach Function With an Intragastric Balloon - a Pilot
Acronym: ANTERO-AC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Prof., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S58484
Record Dates: First submitted 2015-12-08; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Functional Disorders of Stomach

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1. Bag inflated so that intrabagpressure increases with 2 mmHg (Other)
  Interventions: Device: intragastric bag
- 2. Bag inflated to ¾ volume of 1 (Other)
  Interventions: Device: intragastric bag

INTERVENTIONS:
Device: intragastric bag

SUMMARY:
In this pilot study the investigators test the hypothesis that gastric motility can be measured with an intragastric balloon.

ELIGIBILITY:
Inclusion Criteria:

* They are between 18-60 years old.
* Male and female.
* Patients must provide witnessed written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* They are older than 60 years old.
* Have severely decreased kidney function.
* Have severely decreased liver function.
* Have severe heart disease, for example a history of irregular heartbeats, angina or heart attack.
* Have severe lung disease.
* Have severe psychiatric illness or neurological illness.
* Have any gastrointestinal disease.
* Have any dyspeptic symptoms.
* Women that are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Intragastric pressure during food intake | max 3 hours
  The intragastric pressure determined with the manometer and the intragastric bag will be compare before, during and after nutrient drink infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof., Principal Investigator — KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium